CLINICAL TRIAL: NCT00860522
Title: A Phase I Trial of the Immunostimulant JVRS-100 for the Treatment of Patients With Relapsed or Refractory Leukemia
Brief Title: JVRS-100 for the Treatment of Patients With Relapsed or Refractory Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, David F. Claxton, MD, Professor of Medicine, Milton S. Hershey Medical Center
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 08-031
Record Dates: First submitted 2009-03-11; First posted 2009-03-12 (Estimated); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Leukemia
Keywords: relapsed leukemia; refractory leukemia
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phase I (Experimental): Three patients will be enrolled at dose Level 1. If the patient does not completed the three infusion of JVRS-100 during cycle 1 for reason other than toxicity, another patient will be accrued at the same dose level.
  Interventions: Drug: JVRS-100
- Phase II (Experimental): 3 patients will be enrolled at a given dose level. If one of these patients experiences a dose limiting toxicity, an additional 3 patients will be enrolled at the given dose level. If the 1st 2 subjects enrolled and treated at a given dose experience dose limiting toxicities, no additional subjects will be enrolled at that dose. Dose escalation may proceed if < 2/6 patients at a given dose level experience a LDT. If ≥ 2/6 patients experience a DLT at a given dose level, the next lower dose level will be considered the RP2D. If a patient does not complete the 3 infusions of JVRS-100 during Cycle 1 for reasons other than toxicity, another patient will be accrued at the same dose level. Once the RP2D is established, the cohort will be expanded to a total of 12 patients.
  Interventions: Drug: JVRS-100

INTERVENTIONS:
Drug: JVRS-100 — Level 1: 0.5 µg/Kg D1,8,15; Level 2: 1.0 µg/Kg D1,8,15; Level 3:2.0 µg/Kg 1,15; Level 4: 2.0 µg/Kg D1,8,15; Level 5: 4.0 µg/Kg D1,15
  Other Names: Cationic liposome; Plasmid DNA complex
  Arms: Phase I
Drug: JVRS-100 — Change to Stage 2 with starting dose of 4.0 µg/Kg D1,8,15 if no toxicity level by Level 5.
  Other Names: Cationic liposome; Plasmid DNA complex
  Arms: Phase II

SUMMARY:
This is a Phase 1, open-label, dose escalation study of JVRS-100. The study will proceed in 2 stages to minimize the number of patients treated at doses substantially below the recommended phase 2 dose. In stage 1, an accelerated titration schema will be followed with one patient at each dose level. Stage 2 will commence after a dose limiting toxicity is observed in stage 1 or after the maximum dose for stage 1 is reached. Stage 2 will follow a modified Fibonacci schema with 3-6 subjects at each dose level until a recommended phase 2 dose is determined. The cohort will then be expanded to a maximum of 12 patients to more fully evaluate the recommended phase 2 dose.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, dose escalation study of JVRS-100. The study will proceed in 2 stages to minimize the number of patients treated at doses substantially below the recommended phase 2 dose. In stage 1, cohorts of three will be treated at each dose level however doses will be doubled from level to level. Stage 2 will commence after a dose limiting toxicity is observed in stage 1 or after the maximum dose for stage 1 is reached. Stage 2 will follow a modified Fibonacci schema with 3-6 subjects at each dose level until a recommended phase 2 dose is determined. The cohort will then be expanded to a maximum of 12 patients to more fully evaluate the recommended phase 2 dose. The Principal Investigator will assign dose level to be administered to all patients.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* Histologically or cytologically documented relapsed or refractory acute leukemia
* Unlikely to benefit from standard therapy in the opinion of the investigator or refuse standard therapy
* ECOG performance status 0-2
* Adequate renal and hepatic function
* No hematologic criteria for WBC, Hbg or platelets
* Negative virology screen for HIV, hepatitis B surface antigen & hepatitis C
* Female patients of childbearing potential must have a negative serum pregnancy test
* Male & female patients must agree to use a medically acceptable barrier and/or chemical contraceptive method during the study and for a minimum of 3 months afte the last dose of study treatment.
* Patients post blood or marrow transplant should demonstrate a circulating CD8 count of at lest 200 cells/ul

Exclusion Criteria:

* Active CNS leukemia
* Current concomitant chemotherapy, radiation therapy or immunotherapy
* Receipt of any investigational agent within 28 days of first dose of JVRS-100
* Persistent clinically significant toxicity from prior anticancer therapy that is > Grade 2 (NCI CTCAE v3.0)
* Bone marrow or stem cell transplant within 3 months prior to first dose of JVRS-100
* Chronic administration of immunosuppressive agents within 14 days of first dose of JVRS-100. Use of inhaled steroids, nasal sprays, eye drops, and topical creams for small body areas is allowed.
* Pregnant or lactating
* History of prior malignancy other than leukemia within the past 5 years, excluding basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix
* Patients with a systemic fungal, bacterial, viral, or other infection not controlled
* Any condition which, in the opinion of the investigator, would compromise patient safety or compliance, interfere with consent, study participation, follow up, or interpretation of study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-03-01 (Actual); Primary Completion 2014-10-31 (Actual); Study Completion 2017-02-20 (Actual)

PRIMARY OUTCOMES:
Tolerability of JVRS-100 | Day 30 of cycle #1
  Toxicities will be assessed on day 30 of cycle 1. Establish dose limiting toxicity and a maximum tolerated dose recommended Phase 2 dose.

SECONDARY OUTCOMES:
Define parameters of immune activation after JVRS-100 therapy. | Day 30 of cycle #1
  Activation of peripheral blood cells including T-cell subsets, CD4+ and CD8+ cells, B-cells, and NK cells will be studied for activation markers including cell surface phenotypic changes, and expression of intracellular cytokines. Changes in circulating cytokine concentrations will be studied, as will functional properties of circulating immune effector and activating cells.

CONTACTS AND LOCATIONS:
Overall Officials: David F Claxton, MD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Hershey Cancer Institute, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No